CLINICAL TRIAL: NCT02615197
Title: Effectiveness of PTSD Treatment For Suicidal and Multi-Diagnostic Clients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melanie Harned, Research Scientist, Psychology, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49013; R34MH106598 (NIH)
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Post-traumatic Stress Disorder; Suicide; Self-injurious Behavior
Keywords: PTSD; Multi-diagnostic; Dialectical Behavior Therapy; Prolonged Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide; Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical Behavior Therapy (Active Comparator): Standard Dialectical Behavior Therapy (DBT) as described in the 2 DBT treatment manuals (Linehan, 1993; 2014).
  Interventions: Behavioral: Dialectical Behavior Therapy
- Dialectical Behavior Therapy + DBT Prolonged Exposure protocol (Experimental): Standard Dialectical Behavior Therapy (DBT) as described in the 2 DBT treatment manuals (Linehan, 1993; 2014) plus an adapted version of Prolonged Exposure therapy for PTSD.
  Interventions: Behavioral: Dialectical Behavior Therapy; Behavioral: Dialectical Behavior Therapy Prolonged Exposure protocol

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Includes all components of standard DBT (individual therapy, group skills training, phone coaching, and therapist consultation team).
  Other Names: DBT
Behavioral: Dialectical Behavior Therapy Prolonged Exposure protocol — Includes an adapted version of Prolonged Exposure therapy for PTSD.
  Other Names: DBT PE
  Arms: Dialectical Behavior Therapy + DBT Prolonged Exposure protocol

SUMMARY:
The present project has two primary aims: (1) to examine the effectiveness of a multi-component implementation strategy in improving adoption and adherence to the Dialectical Behavior Therapy Prolonged Exposure (DBT PE) protocol, and (2) to evaluate the feasibility, acceptability, and effectiveness of the DBT PE protocol in a sample of individuals receiving DBT in public mental health agencies. This study uses a hybrid type 2 effectiveness-implementation design to simultaneously test the clinical effectiveness of DBT + DBT PE and to evaluate an adaptive, multi-component implementation strategy. The effectiveness trial will use a quasi-experimental, controlled design to evaluate outcomes among DBT clients with PTSD who do versus do not receive the DBT PE protocol and outcomes will be benchmarked to those obtained in research settings.

DETAILED DESCRIPTION:
Although several evidence-based treatments (EBTs) for post-traumatic stress disorder (PTSD) have been found to be effective in research and community settings, individuals with PTSD who are acutely suicidal, self-injuring, and/or have severe comorbid disorders are typically excluded from these treatments. The Dialectical Behavior Therapy Prolonged Exposure (DBT PE) protocol has been shown to be effective in treating PTSD among suicidal, self-injuring, and multi-diagnostic individuals receiving Dialectical Behavior Therapy (DBT) in research settings. The present project has two primary aims: (1) to examine the effectiveness of a multi-component implementation strategy in improving adoption and adherence to the DBT PE protocol, and (2) to evaluate the feasibility, acceptability, and effectiveness of the DBT PE protocol in a sample of individuals receiving DBT in public mental health agencies. The project will be conducted in collaboration with Philadelphia's Department of Behavioral Health and Intellectual disAbility Services (DBHIDS). This study uses a hybrid type 2 effectiveness-implementation design to simultaneously test the clinical effectiveness of DBT + DBT PE and to evaluate an adaptive, multi-component implementation strategy. The effectiveness trial will use a quasi-experimental, controlled design to evaluate outcomes among DBT clients with PTSD who do versus do not receive the DBT PE protocol and outcomes will be benchmarked to those obtained in research settings. Clinical effectiveness outcomes include measures of PTSD, suicidality, global symptom severity, and quality of life and will be assessed at four timepoints (baseline, 4, 8, and 12 months) using blinded independent evaluators. The initial implementation strategy will include an implementation team, online training, distribution of a treatment manual, in-person workshop, team-based clinical consultation, and audit and feedback on session content. The implementation strategy will be adapted as needed during the project using Plan-Do-Study-Act quality improvement methods. Implementation outcomes include feasibility, acceptability, adoption, fidelity, penetration, and sustainability of the DBT PE protocol and will be assessed via clinician surveys at 8 timepoints over 2 years (baseline, pre-training, post-training, 4, 8, and 12-months after initial training during active implementation, and 6 and 12 months follow-up after implementation is complete). Both effectiveness and implementation outcomes are being assessed using mixed methods, including quantitative evaluation (e.g., intent-to-treat analyses across multiple time points) and qualitative evaluation (e.g., surveys and interviews with clients, clinicians, and agency administrators). Four public mental health agencies with existing DBT programs will be recruited for participation. It is estimated that this will yield a sample of 25 clinicians who will enroll a maximum of 3 clients each in the effectiveness trial (n=75 clients total). The project will also engage an advisory board of stakeholders in the DBHIDS system.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for PTSD
* Currently receiving DBT individual therapy with a clinician enrolled in the study

Exclusion Criteria:

* Not able to understand treatment and research assessments conducted in English

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline PTSD Severity at 12 months | Baseline to 12 months
  The PTSD Symptom Scale - Interview will be used to measure the severity of the 17 DSM-IV PTSD symptoms.

SECONDARY OUTCOMES:
Global Severity of Illness | Baseline, 4, 8, and 12 months
  The self-report Brief Symptom Inventory will be used to calculate the Global Severity Index (GSI), which quantifies the patient's overall severity-of-illness.
Health-Related Quality of Life | Baseline, 4, 8, and 12 months
  The self-report CDC Health-Related Quality of Life-4 will be used to assess the number of recent healthy days (i.e., a summary measure of a person's physically and mentally healthy days).
Therapist Adherence to the DBT PE Protocol | Two randomly selected DBT PE therapy sessions per client over the 12 months
  The DBT PE Adherence Scale will be used is an observer-rated measure of the therapist's adherence to the DBT PE protocol during actual therapy sessions.
Mental Health Treatment Utilization | Baseline, 4, 8, and 12 months
  The structured Treatment History Interview will be used to assess utilization of various mental health services (e.g., psychotherapy, psychiatric hospitalization) as well as psychotropic medications.
Intentional Self-Injury | Baseline, 4, 8, and 12 months
  The structured Suicide Attempt Self-Injury Interview will be used to measure the method, intent, medical severity, and outcomes of suicidal and non-suicidal self-injurious behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Harned, PhD, Principal Investigator — University of Washington
Locations (1):
- Behavioral Research and Therapy Clinics, University of Washington, Seattle, Washington, United States